CLINICAL TRIAL: NCT02848768
Title: Validation of a Predictive Nomogram of Response or Resistance to Targeted Therapies in Metastatic Clear Cell Renal Cell Carcinoma
Acronym: RTKI
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_9896
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Sunitinib

SUMMARY:
The purpose of this study is to validate of a predictive nomogram of response or resistance to targeted therapies in metastatic clear cell renal cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* patients with metastatic ccRCC
* Underwent nephrectomy at the University Hospital of Rennes
* treated by sunitinib first line treatment

Exclusion Criteria:

* translocation renal cell carcinoma
* other targeted therapies before the sunitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cohort of 50 patients with metastatic ccRCC who underwent nephrectomy at the University Hospital of Rennes and treated by sunitinib first line treatment.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Primary refractory patients (Progression Free Survival (PFS) | at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France